CLINICAL TRIAL: NCT03908619
Title: A Randomized Controlled Trial of Triple Therapy With Conventional Proton Pump Inhibitor vs Triple Therapy With Vonoprazan as First Line Therapy for Helicobacter Pylori Gastritis
Brief Title: A RCT of Triple Therapy With Proton Pump Inhibitor vs Vonoprazan for Helicobacter Pylori Gastritis
Acronym: TRIVON
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRIVON
Record Dates: First submitted 2019-04-05; First posted 2019-04-09 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori eradication; Triple therapy; Proton pump inhibitor; Vonoprazan
MeSH Terms: interventions — Omeprazole; Esomeprazole; Rabeprazole; 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine

STUDY DESIGN:
Intervention Model Description: Diagnosed H. pylori positive patients (n=252) will be randomized into four study groups:
  * Group A: Omeprazole 20mg bd/ Amoxicillin 1g bd/ Clarithromycin 500mg bd for 14 days (n=42)
  * Group B: Esomperazole 20mg bd/ Amoxicillin 1g bd/ Clarithromycin 500mg bd for 14 days (n=42)
  * Group C: Rabeprazole 20mg bd/ Amoxicillin 1g bd/ Clarithromycin 500mg bd for 14 days(n=42)
  * Group D: Vonoprazan 20mg bd/ Amoxicilllin 1g bd/ Clarithromycin 500mg bd for 7 days (n=42)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TTP (Group A) (Active Comparator): Omeprazole 20mg bd/ Amoxicillin 1g bd/ Clarithromycin 500mg bd for 14 days
  Interventions: Drug: Omeprazole 20mg
- TTP (Group B) (Active Comparator): Esomperazole 20mg bd/ Amoxicillin 1g bd/ Clarithromycin 500mg bd for 14 days
  Interventions: Drug: Esomeprazole 20mg
- TTP (Group C) (Active Comparator): Rabeprazole 20mg bd/ Amoxicillin 1g bd/ Clarithromycin 500mg bd for 14 days
  Interventions: Drug: Rabeprazole Sodium 20mg
- TTP (Group D) (Experimental): Vonoprazan 20mg bd/ Amoxicilllin 1g bd/ Clarithromycin 500mg bd for 7 days
  Interventions: Drug: Vonoprazan

INTERVENTIONS:
Drug: Omeprazole 20mg — Omeprazole 20mg bd/ Amoxicillin 1g bd/ Clarithromycin 500mg bd for 14 days
  Other Names: Losec
  Arms: TTP (Group A)
Drug: Esomeprazole 20mg — Esomperazole 20mg bd/ Amoxicillin 1g bd/ Clarithromycin 500mg bd for 14 days
  Other Names: Nexium
  Arms: TTP (Group B)
Drug: Rabeprazole Sodium 20mg — Rabeprazole 20mg bd/ Amoxicillin 1g bd/ Clarithromycin 500mg bd for 14 days
  Other Names: Pariet
  Arms: TTP (Group C)
Drug: Vonoprazan — Vonoprazan 20mg bd/ Amoxicilllin 1g bd/ Clarithromycin 500mg bd for 7 days
  Other Names: Vocinti
  Arms: TTP (Group D)

SUMMARY:
Helicobacter pylori (H. pylori) gastritis is a common bacterial infection among the elderly population. H. pylori infection causes chronic progressive gastric inflammation, peptic ulcer disease and gastric cancer. Gastric cancer is a significant contributor of cancer-related mortality. The eradication of H. pylori reduces the incidence of gastric cancer. However, the efficacy of H. pylori eradication has decreased dramatically because of antibiotic resistance. This study aims to (i) compare the eradication rates of H. pylori by triple therapy with vonoprazan for the treatment of H. pylori gastritis) (TTV regimen), with triple therapy with conventional proton pump inhibitor (PPI) (TTP regimen) in a multi-racial Asian cohort, (ii) evaluate the prevalence of antibiotic (klacid/amoxicillin/levofloxacin/tetracycline) resistance in H. pylori infected patients, and (iii) assess the safety of the TTV regimen. Diagnosed H. pylori-infected patients (n=252) will be enrolled and randomized 1:1 to TTV or TTP regimen. Gastric biopsies will be cultured and antibiotic sensitivity evaluated using E-test/agar dilution method. The safety of TTV regimen will be assessed using adverse effect questionnaire. This study may potentially impact on prescribing policies and management of H. pylori infections for improved therapeutic outcome.

DETAILED DESCRIPTION:
All subjects who present for endoscopy will be screened. Consent will be taken from subjects who are scheduled to undergo gastroscopy. Gastric biopsies to test for the presence of H. pylori using the rapid CLO test and for culture and sensitivity will be obtained. Based on an estimated prevalence of H. pylori of 20%, we aim to screen approximately 1000 subjects for H. pylori with the rapid CLO test during gastroscopy.

Subjects who have a negative CLO test during endoscopy will be excluded from the study and will be managed accordingly by their physician.

Subjects who are confirmed to have H. pylori gastritis based on the CLO test will then be recruited into the study.

Diagnosed H. pylori positive patients (n=252) will be enrolled into four study groups:

* Group A: Omeprazole 20mg bd/ Amoxicillin 1g bd/ Clarithromycin 500mg bd for 14 days
* Group B: Esomperazole 20mg bd/ Amoxicillin 1g bd/ Clarithromycin 500mg bd for 14 days
* Group C: Rabeprazole 20mg bd/ Amoxicillin 1g bd/ Clarithromycin 500mg bd for 14 days
* Group D: Vonoprazan 20mg bd/ Amoxicilllin 1g bd/ Clarithromycin 500mg bd for 7 days

Randomization codes will be generated by a computer program, and all codes are placed into sealed opaque envelopes and kept by an independent biostatistician. After obtaining informed consent, the investigators would call the research assistant to open the envelope for the allocated regimen. The allocation ratio for TTV and TTP groups is 1:1, with 126 patients in each group. Within the TTP group, the distribution of patients to each of the three PPIs (Omeprazole/Esomeprazole/Rabeprazole) will be equal (n=42 each). The compliance to treatment in terms of percentage of drugs taken will be assessed during clinic review.

This will be a single centre, prospective, open-label, randomized controlled study to (i) compare the eradication rates of H. pylori by TTP regimen vs TTV regimen in a multi-racial Asian cohort, (ii) evaluate the prevalence of antibiotic (clarithromycin/ amoxicillin/ levofloxacin/ tetracycline) resistance in H. pylori-infected patients of both treatment groups, and (iii) assess the safety of the TTV regimen. The proposed study workflow is outlined in Figure 1. This study will be conducted in CGH, in accordance with the ethical principles that have their origin in the Declaration of Helsinki, and are consistent with Good Clinical Practice, applicable regulatory requirements.

The demographic profile (age, gender, ethnicity) and clinical notes (endoscopic findings, antibiotic sensitivity testing results, drug regimen prescribed, extent of treatment compliance, duration of therapy, treatment outcomes i.e. eradication rate, occurrence of adverse events, etc.) of all patients enrolled into the study will be documented for data analysis.

The following experiments will be conducted for the study:

Efficacy assessment:

The success of treatment i.e. eradication of H. pylori is defined as a negative Carbon-13 urea breath test (CUBT) or negative histology test performed at week 6. CUBT or histology will be performed based on the clinical indication as determined by the attending physician. All patients should be off antibiotics and PPI or Vonoprazan for at least 4 weeks prior to assessment of the success of treatment, as per standard practice. All routine laboratory tests will be carried out in Microbiology Lab, Department of Laboratory Medicine, CGH. The technologists will be blinded to the treatment regimens.

Antibiotic susceptibility testing:

For patients with H. pylori infection diagnosed during endoscopy from a positive rapid urease test kit, the material from the test kit will be cultured for antibiotic sensitivity testing. The antibiotic sensitivity testing results may be of value in guiding the choice of antibiotics for second line salvage treatment should first line treatment fails. This has potential usage in the clinical management of patients.

Gastric biopsy specimens collected from both greater gastric corpus and antrum during endoscopy will be inoculated into H. pylori transport medium and transported with ice packs to the laboratory. The biopsy samples will be ground with a tissue homogenizer, cultured, followed by susceptibility testing and determination of the minimum inhibitory concentration (MIC). Briefly, culture will be performed with blood agar medium for Helicobacter with addition of 10% CO2 at 35°C for 7 days. The identity of H. pylori is defined as Gram-negative bacillus with catalase test positive, oxidase test positive, and urease test positive. The MIC of antibiotics (clarithromycin/ amoxicillin/ levofloxacin/ tetracycline) will be determined by E-test or agar plate dilution method in accordance with the guidelines established by the NCCLS Guidelines M100-S9. Mueller-Hinton agar (5% horse blood) will be used with addition of 10% CO2 at 35°C for 72 hours (21). The breakpoint for clarithromycin, amoxicillin, levofloxacin, and tetracycline resistance is defined as ≥ 1.0mg/L, 0.5mg/L, 1mg/L, and 1mg/L, respectively, according to the European Committee on Antimicrobial Susceptibility Testing (EUCAST) (21,22). The laboratory personnel involved in the antibiotic sensitivity testing will be blinded to the study group allocation.

Safety assessment:

An adverse effect questionnaire (AEQ) will be completed by all patients during therapy. The AEQ will contain a checklist to assess the occurrence of loose stools, skin eruption, abdominal bloating, constipation, nausea, epigastric pain, and dysgeusia.

Detection of mutational hotspots for clarithromycin resistance:

An in-house real-time PCR assay will be done on the DNA extracted from the cultured H. pylori isolates to detect mutational hotspots for clarithromycin-resistance.

Post-hoc CYP2C19 genotyping:

Genomic DNA will be extracted from peripheral leukocytes of whole blood using standard desalting methods. Genotyping for the two predominant single nucleotide polymorphisms (CYP2C19*2 and CYP2C19*3) leading to intermediate (heterozygous mutant) and poor metabolizer phenotypes (homozygous mutants) will be performed using sequencing of restriction fragment length polymorphism methods.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed to have H. pylori infection from the Gastroenterology and Hepatology Clinic or ward from Changi General Hospital, The diagnosis of H. pylori infection is established based on either a positive carbon urea breath test (CUBT), a positive rapid urease test, or histology in patients who undergo a diagnostic upper gastrointestinal endoscopy.
* Asian (Chinese, Malay or Indian) ancestry as defined by NRIC,
* Aged ≥ 21 years of age,
* Provision of written informed consent,
* Willing to provide a blood sample for genotyping,
* Ability to communicate with the investigator and to understand and comply with all requirements of study participation.

Exclusion Criteria:

* Known allergy to any of the treatment drugs,
* Inability to undergo routine test to confirm success of H. pylori eradication,
* Previous failed H. pylori therapy,
* Pregnancy or lactation,
* Declare themselves positive for HIV or viral hepatitis (Hepatitis A, B, C),
* Treatment within the previous 3 months with antibiotics.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2019-04-16 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Eradication rates of Helicobacter pylori determined by Carbon-13 urea breath test or biopsy | 6-8 weeks
  Compare eradication rates of Helicobacter pylori by triple therapy with conventional proton pump inhibitor (Omeprazole/ Esomeprazole/ Rabeprazole) (TTP regimen) vs triple therapy with Vonoprazan (TTV regimen) in a multi-racial Asian cohort, using Carbon-13 urea breath test or biopsy

SECONDARY OUTCOMES:
Prevalence of antibiotic resistance based on E-test (Minimum Inhibitory Concentrations) | 6-8 weeks
  Evaluate the prevalence of antibiotic (clarithromycin/ amoxicillin/ levofloxacin/ tetracycline) resistance in H. pylori-infected patients of both treatment groups using E-test
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 8 weeks
  Assess the safety of triple therapy for eradication of H. pylori in the local population using adverse effect questionnaire
Association of CYP2C19 genotypes with triple therapy efficacy | Through study completion, an average of 2 years
  Perform CYP2C19 using sequencing or restriction fragment length polymorphism methods

CONTACTS AND LOCATIONS:
Overall Officials: Daphne Shih Wen Ang, MD, Principal Investigator — Changi General Hospital
Locations (1):
- Clinical Trials & Research Unit, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li M, Oshima T, Horikawa T, Tozawa K, Tomita T, Fukui H, Watari J, Miwa H. Systematic review with meta-analysis: Vonoprazan, a potent acid blocker, is superior to proton-pump inhibitors for eradication of clarithromycin-resistant strains of Helicobacter pylori. Helicobacter. 2018 Aug;23(4):e12495. doi: 10.1111/hel.12495. Epub 2018 Jun 6. PMID 29873436
- [Background] Sue S, Kuwashima H, Iwata Y, Oka H, Arima I, Fukuchi T, Sanga K, Inokuchi Y, Ishii Y, Kanno M, Terada M, Amano H, Naito M, Iwase S, Okazaki H, Komatsu K, Kokawa A, Kawana I, Morimoto M, Saito T, Kunishi Y, Ikeda A, Takahashi D, Miwa H, Sasaki T, Tamura T, Kondo M, Shibata W, Maeda S. The Superiority of Vonoprazan-based First-line Triple Therapy with Clarithromycin: A Prospective Multi-center Cohort Study on Helicobacter pylori Eradication. Intern Med. 2017;56(11):1277-1285. doi: 10.2169/internalmedicine.56.7833. Epub 2017 Jun 1. PMID 28566587